CLINICAL TRIAL: NCT04471909
Title: A Multi-arm, Multi-Center, Non-Randomized, Prospective, Clinical Study to Evaluate the Safety and Effectiveness of the NEXUS Aortic Arch Stent Graft System in Treating Thoracic Aortic Lesions Involving the Aortic Arch
Brief Title: NEXUS Aortic Arch Clinical Study to Evaluate Safety and Effectiveness
Acronym: TRIOMPHE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Endospan Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-009
Record Dates: First submitted 2020-07-09; First posted 2020-07-15 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Aortic Dissection; Aortic Aneurysm; Intramural Hematoma; Penetrating Aortic Ulcer
MeSH Terms: conditions — Aortic Dissection; Aortic Aneurysm; Penetrating Atherosclerotic Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Chronic Dissection (arm closed to enrollment) (Experimental)
  Interventions: Device: NEXUS Aortic Stent Graft System
- Penetrating Aortic Ulcer and/or Intramural Hematoma (Experimental)
  Interventions: Device: NEXUS Aortic Stent Graft System
- Aneurysm (arm closed to enrollment) (Experimental)
  Interventions: Device: NEXUS Aortic Stent Graft System

INTERVENTIONS:
Device: NEXUS Aortic Stent Graft System — Arch Stent Graft, whose cranial narrow end is intended to be deployed into the Brachiocephalic artery and whose distal end is intended to be deployed into the Descending Thoracic Aorta.
  Ascending Stent Graft intended to be deployed in the Ascending Aorta.
  OPTIONAL: Descending Extension can be used in case the aortic lesion elongates further distally and out of the covered length offered by the Arch Stent Graft. Multiple Descending Extensions can be used if needed to cover the entire length of the lesion.

SUMMARY:
Prospective, non-randomized, multi-center clinical investigation of the NEXUS™ Aortic Arch Stent Graft System (NEXUSTM) for the treatment of thoracic aortic lesions involving the aortic arch with a proximal landing zone, native or previously implanted surgical graft, in the ascending aorta and with a brachiocephalic trunk native landing zone.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female age ≥ 18.
2. Proximal/ascending native or previously implanted surgical graft landing zone of appropriate length
3. Proximal/ascending native or previously implanted surgical graft landing zone of appropriate diameter
4. Distal/descending native landing zone of appropriate length
5. Distal/descending native landing zone of appropriate diameter
6. Brachiocephalic trunk native landing zone of appropriate length
7. Brachiocephalic trunk native landing zone of appropriate diameter
8. Appropriate take off angle between the Brachiocephalic Artery and the Aortic Arch perpendicular
9. Appropriate aortic arch perpendicular diameter
10. Chronic dissection with at least one of the following conditions:

    1. An aortic aneurysm with a maximum diameter ≥ 55 mm
    2. Rapidly expanding false lumen (growth of > 0.5 cm/6 months)
    3. Compressed true lumen associated with end organ malperfusion
    4. Symptomatic
11. Aneurysm with at least one of the following conditions:

    1. Dilatation of the aortic arch larger than 5 cm in diameter for subject with fusiform aneurysm
    2. Dilatation of the aortic arch is 1.5 times the normal diameter for subjects ascending or descending
    3. Dilation of the aortic arch larger than 2.5 cm for subject with saccular aneurysm
    4. Symptomatic aneurysm of the aortic arch
    5. Aortic diameter growth rate > 5mm per 6 months
    6. Postoperative pseudoaneurysm expanding from anastomotic suture lines
12. Penetrating aortic ulcer with at least one of the following:

    1. Symptomatic
    2. Ulcer demonstrates expansion
13. Intramural hematoma with at least one of the following:

    1. Symptomatic (persistent pain)
    2. Transverse or longitudinal expansion on serial imaging
14. In the event of a lesion in the ascending aortic, the proximal/ascending native or previously implanted surgical graft the landing zone must be appropriate
15. Femoral / iliac artery diameter as documented by CTA or MRA that allows endovascular access to the diseased site with a 20 Fr. delivery catheter.
16. Access vessels morphology suitable for endovascular repair in terms of tortuosity, calcification and angulation, documented by CTA/MRA.
17. Brachial/Axial Artery diameter that allows endovascular access suitable for 7 Fr.
18. Subject is considered an appropriate candidate for an elective surgery.
19. Subject is considered to be at high risk for open repair, as determined by the investigator.
20. Access vessels, iliac/femoral & brachial/axillary compatible with vascular access techniques (femoral cutdown or percutaneous), devices, and /or accessories.
21. Subject is willing and able to comply with procedures specified in the protocol and is able to return for follow-up visits as specified by the protocol.

Exclusion Criteria:

1. Acute dissection
2. Lesions that can be safely treated with TEVAR landing in zone 2 (with or w/o LSA vascularization)
3. Required emergent treatment, e.g., trauma, rupture
4. Acute vascular injury of the aorta due to trauma
5. Aortic rupture or unstable aneurysm
6. Received a previous stent or stent graft in the treated area (including planned landing area)
7. Required surgical or endovascular treatment of an infra-renal aneurysm at time of implantation
8. Planned major surgical or interventional procedure at time of screening, to be performed after the NEXUS™ implantation.
9. Any major surgical or interventional procedure 6 weeks before the NEXUS™ implantation, exclusive of planned procedures that are needed for the safe and effective placement of the stent graft (e.g. supra-aortic bypass).
10. Subject has had a myocardial infarction (MI) or cerebral vascular accident (CVA) within 90 days prior to the planned implantation
11. Subjects with severe aortic valvular insufficiency as determined by echocardiography
12. Mechanical valve that preclude safe delivery of NEXUS™
13. Known Connective tissue disease (e.g., Marfan's or Ehler's-Danlos syndromes)
14. Subject has an active systemic infection at the time of the procedure documented by pain, fever, drainage, positive culture
15. Pregnant
16. Life expectancy of less than 2 years
17. Unsuitable vascular anatomy
18. Subject who have a previously implanted surgical wrap of the ascending aorta
19. Any medical condition that, according to the investigator's decision, might expose the subject to increased risk by the investigational device or procedure.
20. An aneurysm that is mycotic, inflammatory or suspected to be infected.
21. Subject with hostile groins/axilla (scarring, obesity, or previous failed puncture) unless conduit are used.
22. Subjects with severe atherosclerosis, severe calcification or extensive intraluminal thrombus of the aorta or in the brachiocephalic trunk
23. Subject is suffering from unstable angina or NYHA classification III and IV.
24. Subject has a known hypersensitivity or contraindication to anticoagulants, antiplatelets, or contrast media, which is not amenable to pre-treatment.
25. Subject with a contraindication to undergo angiography
26. Subject with known sensitivities or allergies to the device materials (including Nitinol [NiTi], polyester fabric [PET], tantalum [TA])
27. Clinical conditions that severely inhibit x-ray visualization of the Aorta.
28. Subject has history of bleeding diathesis or coagulopathy that may limit the use of dual antiplatelet or anticoagulant therapy by the decision of the investigator
29. Acute renal failure; chronic renal failure (excluding dialysis); Creatinine > 2.00 mg/dl
30. Any other medical, social, or psychological issues that in the opinion of the investigator preclude them from receiving this treatment, or the procedures and evaluations pre- and post- treatment.
31. Active participation in another clinical study that has not completed primary endpoint(s) evaluation or that clinically interferes with the endpoints in this study, or subject is planning to participate in such study prior to the completion of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2020-10-20 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Device Technical Failure | 30 Days
  * Failure to accurately deliver, track and deploy all required endovascular device components at the intended implantation site and failure to retrieve the device delivery systems without the need for unplanned additional procedures
  * Device occlusion
  * Failed exclusion of primary entry tear
  * Additional unanticipated surgical or interventional procedure related to the device or procedure, to prevent life-threatening or permanent disabling event.
Clinical Failure | 30 Days
  Subjects experiencing early mortality or at least one of the following MAEs through 30-Day of Phase 1 Procedure and 30-Day of Index Procedure: Disabling stroke, permanent paralysis/paraplegia, renal failure, aortic rupture, development of new dissections in the thoracic aorta or brachiocephalic artery.

CONTACTS AND LOCATIONS:
Locations (32):
- United States (31):
  - University of Alabama Birmingham, Birmingham, Alabama
  - University of California San Diego Medical Center, La Jolla, California
  - UC Davis Health, Sacramento, California
  - Stanford University School of Medicine, Stanford, California
  - University of Colorado, Aurora, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - MedStar Washington Hospital, Washington D.C., District of Columbia
  - Advent Health Orlando, Orlando, Florida
  - Emory University, Atlanta, Georgia
  - The University of Chicago, Chicago, Illinois
  - Ascension St. Vincent, Carmel, Indiana
  - University of Maryland, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - The Mount Sinai Medical Center, New York, New York
  - Northwell Health Lenox Hill Hospital, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Atrium Health, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - The Lindner Research Center, Cincinnati, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Oregon Health, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Ballad Health, Kingsport, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor Scott and White, Plano, Texas
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Carilion Clinic, Roanoke, Virginia
- Auckland City Hospital, Auckland, Grafton, New Zealand